CLINICAL TRIAL: NCT05734508
Title: Cohort Events Monitoring (CEM) Study for the Assessment of Safety Profile of MVA-BN (Jynneos) Vaccine in Adult Personnel and Staff in the PALM-007 Study in Democratic Republic Of The Congo
Brief Title: Assessment of Safety Profile of MVA-BN Vaccine in the PALM-007 Study in DRC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PALM 008
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MVA-BN vaccine (Experimental): 2 doses of 0.5 mL MVA-BN vaccine injected subcutaneously and given at least 28 days apart
  Interventions: Biological: MVA-BN vaccine

INTERVENTIONS:
Biological: MVA-BN vaccine — A live vaccine produced from the Modified Vaccinia Ankara-Bavarian Nordic strain (MVA-BN), an attenuated and non-replicating orthopox virus
  Other Names: JYNNEOS

SUMMARY:
The goal of this observational study is to monitor and assess the safety profile of the MVA-BN vaccine among staff and study personnel of the PALM-007 study in the Democratic Republic of the Congo. The main questions it aims to answer are:

* To estimate the incidence of serious adverse events (SAEs) in all individuals vaccinated with the MVA-BN vaccine
* To estimate the incidence of adverse events (AEs) after each dose of MVA-BN vaccine.

Participants will receive two doses of vaccine and will be actively followed up to the 28th day after their last dose of MVA-BN vaccine.

DETAILED DESCRIPTION:
All personnel and staff of the PALM-007 study will be offered the opportunity to participate in the study by reviewing and signing the informed consent. After signing informed consent, participants will be examined. The following parameters will be assessed:

* Anthropometric measurements (weight, height)
* Vital signs: temperature (axillary), blood pressure, heart rate and respiratory rate
* Medical history, including history of orthopox virus disease, vaccination, current co-morbidities and medication(s)
* Physical examination
* Pregnancy test will be done for all women of childbearing potential

If a participant has met all eligibility criteria, they will be enrolled and will receive the vaccine as specified below. Participants who are excluded because of fever can be rescreened and included after resolution of the fever and its cause.

Enrolled participants will receive the MVA-BN vaccine by subcutaneous injection of 0.5 mL in the shoulder (left or right).

The first dose will be administered at the time of enrollment and the second dose 28 days later.

After each vaccination, the participant will remain under observation for 30 minutes. All AEs occurring during this period of observation will be recorded and reported to the National Center for Pharmacovigilance and to the ethics committee according to Congolese regulations.

Follow-up of participants:

Participants will be followed until 28 days after the second dose of vaccine. Follow-up visit will be done either in person at National Institute of Biomedical Research (INRB) in Kinshasa and at the Monkeypox treatment centers in the PALM-007 study or by phone calls on Day 3, Day 14, and Day 28 post each vaccination. Study participants will be provided with contact information of vaccine research staff and have the right to contact the research team either directly or by phone if they have any questions about post-vaccination reactions they may be experiencing or if they are concerned. There is a window of +/- one day for each study visit except the day of the second dose which can be done on day 28 after the first dose with a window of +7 days. This second dose must not be given before Day 28. During each visit, participants will be asked to report to the research team AEs via open-ended questions. All SAEs will be followed-up. SAEs that have not resolved by the end of the per-protocol follow-up period for the subject (Day 28 after second dose) are to be followed until final outcome is known (to the degree permitted by the IRB-approved informed consent form). If it is not possible to obtain a final outcome for an SAE (e.g., the participant is lost to follow-up), the last known status and the reason a final outcome could not be obtained will be recorded by the investigator on an SAE report update and the CRF.

On the day of administration of the second dose of vaccine, vital signs, and physical examination will be done to all participants and a pregnancy test will be done on all women of childbearing potential prior to vaccine administration. If the pregnancy test is positive, the second dose will not be given, and the participant will be followed up as described in the protocol. Participants will be instructed to report any AEs that are experienced outside of the protocol defined follow up days. The reporting form of the national pharmacovigilance system of the DRC will be used for reporting. The research team will complete the notification form which will be sent to the National Pharmacovigilance Center (CNPV) by e-mail (scanned copies).

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent
* 18 years of age or older
* At high risk for Monkeypox infections
* Personnel and staff associated with the PALM 007-Monkeypox study sites in the DRC
* Willingness and ability to communicate AEs to study personnel

Exclusion Criteria:

* Allergy to MVA-BN or any of its components
* Pregnant or breastfeeding women
* Fever (axillary temperature ≥37.5°celsius)
* People who have already received the MVA-BN vaccine (in routine vaccination or another study involving this vaccine)
* Participants who, in the judgement of the investigator, will be at significantly increased risk as a result of participation in the study
* Individuals with any condition or circumstance that would render them unable to comply with study procedures (e.g., not reachable by phone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Democratic Republic of the Congo (3):
  - Institut National de Rescherche Biomédicale (INRB), Kinshasa
  - L'Hôpital Général de Référence de Kole, Kole
  - L'Hôpital Général de Référence de Tunda, Tunda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at three sites from March 2023 to June 2024. The first two sites were Tunda and Kole General Hospitals, in Maniema and Sankuru provinces, DRC (the two sites where participants with mpox were enrolled in the PALM 007 therapeutic RCT). The third site subsequently opened at the INRB main campus in Kinshasa, DRC. Adult participants (≥18 years) were recruited from PALM 007 study staff, although it was not mandatory for staff to be vaccinated or participate in the trial.
Groups:
- MVA-BN Mpox Vaccine: This arm, which includes all participants in this observational safety study, received the Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN) vaccine, an attenuated, live, non-replicating virus, administered in two doses separated by at least 28 days.
Period: Overall Study
Arm/Group | MVA-BN Mpox Vaccine
Started | 500
Received First Vaccine Dose | 500
Received Second Vaccine Dose | 494
Completed | 494
Not Completed | 6
Not completed — Pregnancy | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | MVA-BN Mpox Vaccine
Number analyzed (Participants) | 500
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 391
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Frequency of SAEs After First Dose of MVA-BN Vaccine
Description: Number of participants with an SAE up to 14 days after dose
Time Frame: Within 14 days of first vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN Mpox Vaccine
Number analyzed (Participants) | 500
Participants | 0

2. Primary Outcome: Frequency of SAEs After Second Dose of MVA-BN Vaccine
Description: Number of participants with an SAE up to 14 days after dose
Time Frame: Within 14 days of second vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN Mpox Vaccine
Number analyzed (Participants) | 494
Participants | 0

3. Primary Outcome: Frequency of AEs After First Dose of MVA-BN Vaccine
Description: Number of participants with an AE within 14 days of first vaccine dose
Time Frame: Within 14 days of first vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN Mpox Vaccine
Number analyzed (Participants) | 500
Participants | 219

4. Primary Outcome: Frequency of AEs After Second MVA-BN Vaccine Dose
Description: Number of participants with an AE up to 28 days after second vaccine dose
Time Frame: Within 28 days of second vaccine dose
Measure: Count of Participants; unit: Participants
Arm/Group | MVA-BN Mpox Vaccine
Number analyzed (Participants) | 494
Participants | 102

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 28 days after receipt of the second vaccine dose
Arm/Group | MVA-BN Mpox Vaccine
All-Cause Mortality (participants affected / at risk) | 0/500
Serious Adverse Events (participants affected / at risk) | 0/500
Other Adverse Events (participants affected / at risk) | 281/500
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MVA-BN Mpox Vaccine (N=500)
Pyrexia (General disorders and administration site conditions) | 67 (67)
Vaccination site pain (General disorders and administration site conditions) | 164 (164)
Headache (Nervous system disorders) | 72 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT05734508/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT05734508/ICF_001.pdf